CLINICAL TRIAL: NCT06695598
Title: An Open Label, Randomized, Single Dose, Crossover, Phase I Study to Evaluate the Effects of Food on Pharmacokinetics and the Safety of CKD-383 in Healthy Adult Volunteers
Brief Title: Clinical Study to Evaluate the Food Effect of CKD-383 0.5/25/1000mg in Healthy Volunteers
Acronym: CKD-383 FDI P1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A101_08FDI2414
Record Dates: First submitted 2024-11-17; First posted 2024-11-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fast-Fed (Experimental): Period 1: A single oral dose of 1 tablet under fasting condition, Period 2: A single oral dose of 1 tablet under fed condition
  Interventions: Drug: CKD-383
- Fed-Fast (Experimental): Period 1: A single oral dose of 1 tablet under fed condition, Period 2: A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-383

INTERVENTIONS:
Drug: CKD-383 — QD, PO

SUMMARY:
This study is a randomized, open-label, single dose, crossover study to evaluate the food effect of CKD-383 in healthy volunteers

DETAILED DESCRIPTION:
To 30 healthy subjects, following treatments are administered dosing in each period and wash-out period is 7 days

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults volunteers between the ages of 19 years to 55 years.
2. Individuals who had 18.0 kg/m2 ≤ Body Mass Index(BMI) < 30.0 kg/m2 and total body weight ≥ 50 kg (woman total body weight ≥ 45 kg) BMI = Weight(kg)/ Height(m)2
3. Following vital signs results at screening

   * Systolic blood pressure: 90 mmHg to 150 mmHg
   * Diastolic blood pressure: 50 mmHg to 100 mmHg
4. Individuals who is determined by investigators to be suitable as a test subject as a result of the examination conducted at the time of screening
5. Individuals who agreed proper contraception during the study and did consent to not donation of sperm 7 days after the last dose of study drug
6. Individuals who signed an informed consent form after being fully informed of the study prior to participation, including the objective and content

Exclusion Criteria:

1. Clinically significant biliary tract (such as hepatic dysfunction, liver failure, etc.), kidney (stage 3b), and severe renal impairment (eGFR <60 mL/min/1.73 m2), nervous system, immune system, respiratory system (such as pulmonary infarction, severe pulmonary dysfunction and other hypoxemia prone conditions, respiratory failure, etc.), urinary system, digestive system (such as diarrhea and vomiting), endocrine system, blood and tumor, cardiovascular system (acute myocardial infarction, shock, acute and unstable heart failure, decompensated heart failure, severe heart failure, or those with a history of heart failure (such as New York Heart Association(NYHA) Classification 3 and 4 heart failure)
2. Acute or chronic metabolic acid patients with type 1 diabetes, lactic acidosis, diabetic ketoacidosis with or without a coma, and diabetic ketoacidosis patients
3. Patients with diabetic comas and ex-marriage
4. Individuals who have an acute condition that can change his or her renal function, such as dehydration, before and after surgery, severe infection, severe traumatic systemic disorder, cardiovascular collapse (shock), sepsis, etc
5. Patients undergoing intravenous examination of radiodine contrast agents (e.g., intravenous urinary tract, intravenous cholangiography, angiography, computed tomography with contrast agents, etc.)
6. Patients with malnutrition, starvation, weakness, pituitary dysfunction or adrenal insufficiency
7. Individuals who have a history of gastrointestinal diseases (Cron's disease, ulcerative colitis, etc.) or surgery (excluding simple appendectomy or hernia surgery) that may affect the absorption of drugs
8. Individuals who have a history of clinically significant hypersensitivity reactions to the main components and components of clinical trial drugs and other drugs (viguanide drugs, thiazolidinedione drugs, etc.)
9. Individuals who have a history of drug abuse within one year of screening or who has tested positive for a urine drug test
10. Pregnant women, women who may be pregnant, nursing women
11. Those who consumed excessive smoking or caffeine or alcohol within one month prior to the first administration of clinical trial drugs (caffeine: >5 cups/day, alcohol: male: >21 cups/week, female: >14 cups/week, tobacco: >20 cigarettes/day), or who cannot stop smoking, caffeine and alcohol consumption during each hospitalization period
12. If the investigators determines that the drug may affect the clinical trial or the safety of the subject by administering prescription drugs or herbal medicines within 14 days prior to the first administration of investigational product or general medicines including health foods and vitamin preparations within 7 days
13. Individuals who have taken a drug metabolase-inducing and inhibiting drug, such as barbitals, within 30 days prior to the first administration of investigational product
14. Individuals who had been administered investigational product from other clinical study(include bioequivalence study) within the 6 months prior to the first administration of investigational drugs
15. Individuals who donated whole blood within the 8 weeks, or blood components within 2 weeks or had a blood transfusion within 30 days prior to the first administration of investigational drugs
16. Those who are deemed insufficient to participate in this clinical study by investigators

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-383 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hours
  Area under the CKD-383 concentration in blood-time curve from 0 to t
Cmax of CKD-383 | 0, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48 hours
  The maximum CKD-383 concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Locations (1):
- Bumin Hospital, Gangseo-gu, Seoul, South Korea